CLINICAL TRIAL: NCT01843140
Title: Fertility Information Research Study
Brief Title: Assessing Reproductive Outcomes in Young Female Cancer Survivors Through a National Fertility Preservation Registry
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Hui-Chun Irene Su, Assistant Professor of Reproductive Medicine, University of California, San Diego
Other Study IDs: FIRST
Record Dates: First submitted 2012-07-26; First posted 2013-04-30 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Cancer; Infertilty
Keywords: cancer; fertility preservation; infertility; pregnancy
MeSH Terms: conditions — Neoplasms; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dried blood spots
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Young female cancer survivors

SUMMARY:
The FIRST project is a national fertility preservation registry for young women facing cancer treatments. The investigators will examine how different cancers and treatments affect the reproductive health of young survivors. This prospective cohort study seeks to recruit young women close to time of cancer diagnosis and treatment. Participants will answer a yearly questionnaire on their current health. A subset of participants will provide dried blood spots to measure reproductive hormones. The primary goal of the study is to determine the risk of infertility and time to pregnancy in young female cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer or exposure to cancer treatment
* English speaking
* Ability to consent to the study

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young women ages 18-44 who have been diagnosed with cancer or exposed to cancer treatment
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Risk of infertility | Annually up to 10 years
  Participants will be assessed for infertility on average each year from age 18 to 51, the age of natural menopause.

SECONDARY OUTCOMES:
Time to pregnancy | Annually up to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

REFERENCES:
- [Derived] Dominick SA, McLean MR, Whitcomb BW, Gorman JR, Mersereau JE, Bouknight JM, Su HI. Contraceptive Practices Among Female Cancer Survivors of Reproductive Age. Obstet Gynecol. 2015 Sep;126(3):498-507. doi: 10.1097/AOG.0000000000000963. PMID 26181090